CLINICAL TRIAL: NCT01844375
Title: A Randomized Controlled Trial of Preoperative Carbohydrate Drinks on Postoperative Walking Capacity in Colorectal Surgery.
Brief Title: A Trial of Preoperative CHO Drinks on Postoperative Walking Capacity in Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mingkwan Wongyingsinn, MD (Other)
Responsible Party: Sponsor-Investigator, Mingkwan Wongyingsinn, MD, Assistant professor, Doctor, Siriraj Hospital
Organization: Siriraj Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SIRB050
Record Dates: First submitted 2013-04-22; First posted 2013-05-01 (Estimated); Results first posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Bowel; Disease, Carbohydrate Absorption; Difficulty Walking; Colorectal Neoplasms
Keywords: oral carbohydrate loading; walking capacity
MeSH Terms: conditions — Disease; Mobility Limitation; Colorectal Neoplasms | interventions — Control Groups; Water

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carbohydrate group (Experimental): The carbohydrate (CHO) group will be given the carbohydrate drink (12.5% carbohydrates, 50 kcal/100 ml, 240 mOsmol/l, pH 5.0) 800 mL of one of the drinks the night before surgery, between 1900 and 2400 h, and another 400 ml in the morning of the operation day. The last drink will be no later than 3 hours before the scheduled induction of anesthesia. Of note, the last meal on the day before the operation will be no later than 1800 h. Following this meal, no food or drink will be allowed except the carbohydrate drink. The pharmacy department is responsible for preparing the carbohydrate drink.
  Interventions: Dietary Supplement: Carbohydrate group
- Control group (Active Comparator): The control group will be given pure water 800 mL of one of the drinks the night before surgery, between 1900 and 2400 h, and another 400 ml in the morning of the operation day. The last drink will be no later than 3 hours before the scheduled induction of anesthesia. Of note, the last meal on the day before the operation will be no later than 1800 h. Following this meal, no food or drink will be allowed except pure water.
  Interventions: Other: Control group

INTERVENTIONS:
Dietary Supplement: Carbohydrate group — The patients will be given 12.5% carbohydrates drink 800 mL the night before surgery, between 1900 and 2400 h, and another 400 ml in the morning.
  Other Names: carbohydrate drink; carbohydrate supplement
  Arms: Carbohydrate group
Other: Control group — The patients will be given water 800 mL to drink the night before surgery, between 1900 and 2400 h, and another 400 ml in the morning.
  Other Names: pure water; water
  Arms: Control group

SUMMARY:
This prospective randomized controlled study is designed to investigate whether preoperative oral carbohydrate loading improves postoperative walking performance, a surrogate indicator for overall functional recovery, in patients undergoing colorectal surgery as measured by 2-minute and 6-minute walk test. The secondary outcomes are postoperative insulin resistance measured with plasma insulin and glucose concentrations. The tertiary outcomes are duration of hospital stay, patients satisfaction during staying in the hospital and morbidity measured as postoperative complications.

DETAILED DESCRIPTION:
After approval by the Siriraj Institutional Review Board, patients aged greater than 18 years undergoing elective colorectal surgery at Siriraj Hospital will be approached and recruited in this study. Exclusion criteria are diabetes mellitus, any endocrine disorders or metabolic abnormalities, impaired renal function (GFR <60 ml/min), impaired hepatic function (Child-Pugh score class C), a history of delayed gastric emptying time, body mass index >30, inability to communicate and severe physical disability. Informed written consent will be obtained from each subject.

At the time of admission to the hospital, patients will be randomly allocated to one of the two groups using a computer-generated randomization schedule in a block of five. The carbohydrate (CHO) group will be given the carbohydrate drink (12.5% carbohydrates, 50 kcal/100 ml, 240 mOsmol/l, pH 5.0) while the control group will be given pure water. The pharmacy department is responsible for preparing the carbohydrate drink. The patients in the two groups will be given 800 mL of one of the drinks the night before surgery, between 1900 and 2400 h, and another 400 ml in the morning of the operation day. The last drink will be no later than 3 hours before the scheduled induction of anesthesia. Of note, the last meal on the day before the operation will be no later than 1800 h. Following this meal, no food or drink will be allowed except the carbohydrate drink or pure water.

Before induction of anesthesia, a thoracic epidural catheter will be inserted as routine in either the ninth or tenth thoracic intervertebral space in patients undergoing laparotomy colorectal surgery. Lidocaine 2% with epinephrine 1:200,000 3 mL will be injected in the epidural space to produce a bilateral segmental sensory block to ice and pinprick between T6 and T12 dermatomes. The neural blockade was maintained during surgery with additional infusion of bupivacaine 0.25% 4-8 mL/h.

General anesthesia will be induced in all patients with same protocol. Preoperative mechanical bowel preparation will be utilized in the case of left-sided colon cancer or rectal cancer. Intravenous prophylactic antibiotics will be administered to every patient. All operations will be performed by well-experienced surgeons. The choice of incision and operation will depend on tumor location and surgeon's discretion.

Primary outcomes are 2-minute walk test (2MWT) which will be measured before surgery to be a baseline, and then 2MWT will be measured at 72 hours after surgery. Patients will be asked to walk back and forth along a 15 m stretch of hallway as much as they can over a period of 2 minutes. To ensure safety, the evaluator walks behind the patient. Patients are told that they can rest if necessary, and they are allowed to use their regular walking aids.

Serum insulin and glucose concentrations will be measured preoperatively, and on the first three postoperative days. Blood sample for insulin will be centrifuged (Cobas® 8000 modular analyzer series; modular pre-analytics evo, Roche) at 3000 rpm for 5 min at 22.5°C and insulin level will be measured by a two-site immunoassay using electrochemiluminescence immunoassay (ECLIA) (Cobas® 8000 modular analyzer series: e 602 module, Roche). Blood sample for glucose will be immediately centrifuged (Kokusan H-28F, Euroscan) at 3500 rpm for 10 min at 25°C and glucose concentration will be measured using an enzymatic (Hexokinase) method (Cobas integra® 800 analyzer; c 702 module, Roche).

24-Hour urine urea nitrogen will be measured on the first three postoperative days. The urine sample will be centrifuged (Cobas® 8000 modular analyzer series; modular pre-analytics evo, Roche) at 3000 rpm for 5 min at 22.5°C and measured using a urease/glutamate dehydrogenase coupled enzymatic technique (Cobas 8000 modular analyzer series: c 702 module, Roche).

Postoperative pain at rest and on mobilization at postoperative 24, 48 and 72 hours will be assessed with verbal rating score (VRS) from 0 (no pain) to 10 (worst pain). Postoperative use of analgesics and amount of analgesic medication will be recorded daily during the first three postoperative days. The duration of hospital stay will be measured by time (days) from the day of surgery to the day of discharge. Patient satisfaction during staying in the hospital will be assessed when discharging from the hospital with a verbal rating score

ELIGIBILITY:
Inclusion Criteria:

- patients aged greater than 18 years undergoing elective colorectal surgery at Siriraj Hospital

Exclusion Criteria:

* diabetes mellitus
* any endocrine disorders or metabolic abnormalities
* impaired renal function (GFR <60 ml/min)
* impaired hepatic function (Child-Pugh score class C)
* a history of delayed gastric emptying time
* body mass index >30
* inability to communicate
* severe physical disability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mingkwan Wongyingsinn, MD, MSc, Study Director — Siriraj Hospital
Locations (1):
- Siriraj hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Carbohydrate Group | Control Group
Started | 35 | 35
Completed | 34 | 34
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carbohydrate Group | Control Group | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (10.2) | 62.7 (9.7) | 62.8 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 13 | 30
  Male | 17 | 21 | 38
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 22.1 (3.1) | 23.2 (3.9) | 22.6 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: Meters Walked During 2-Minute Walk Test
Description: Primary outcomes are 2-minute walk test (2MWT) which will be measured before surgery to be a baseline, and then 2MWT will be measured at 72 hours after surgery. Patients will be asked to walk back and forth along a 15 m stretch of hallway as much as they can over a period of 2 minutes. To ensure safety, the evaluator walks behind the patient. Patients are told that they can rest if necessary, and they are allowed to use their regular walking aids. Any intravenous lines, tubes, or infusion pumps will be attached to a pole and pushed by the patient. The walking distance will be recorded in meters. If the patient is unwilling or unable to walk, the reason will be recorded and the distance '0' will be recorded for that day.
Time Frame: 72 hours after surgery
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Carbohydrate Group | Control Group
Number analyzed (Participants) | 34 | 34
meters | 70 [48 to 102] | 64 [55 to 94]
Statistical Analysis 1: Comparison: Carbohydrate Group vs Control Group; Test type: Equivalence — equivalence analysis; p = 0.75, Kruskal-Wallis

2. Secondary Outcome: Change of Serum Glucose Concentration
Description: Serum glucose concentrations will be measured preoperatively, and on the 24 hour postoperatively.
Time Frame: Baseline and postoperative 24 hours
Measure: Median (Inter-Quartile Range); unit: microunit/mL
Arm/Group | Carbohydrate Group | Control Group
Number analyzed (Participants) | 34 | 34
microunit/mL | 3.2 [-7.1 to 11.9] | 3.8 [-3.5 to 8.2]

3. Secondary Outcome: Nitrogen Balance
Description: 24-hour urine urea nitrogen was measured on the postoperative day 3.
  The urine samples during 24 hours on the postoperative day 3 were centrifuged (Cobas 8000 Modular Analyzer Series; Modular Pre-analytics Evo, Roche) at 3000 rpm for 5 min at 22.5°C, and measured using a urease/glutamate dehydrogenase coupled enzymatic technique (Cobas 8000 Modular Analyzer Series: C 702 Module, Roche). The nitrogen balance was calculated by measuring urinary urea nitrogen and dietary nitrogen intake during the same 24-hour period. The nitrogen intake was estimated for each patient following a doctor's diet order and types of food formulas in hospital, and then dividing the daily protein intake by 6.25. The urine urea nitrogen was added by 4 to account for non-urinary losses of nitrogen
Time Frame: on the postoperative day 3
Measure: Median (Inter-Quartile Range); unit: mg/mL
Arm/Group | Carbohydrate Group | Control Group
Number analyzed (Participants) | 34 | 34
mg/mL | 4.7 [2.9 to 6.3] | 3.1 [-4.8 to 5.3]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Carbohydrate Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 6/34 | 4/34
Other Adverse Events (participants affected / at risk) | 0/34 | 0/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carbohydrate Group (N=34) | Control Group (N=34)
Infected surgical wound (Infections and infestations) | 2 (2) | 2 (2)
Bowel ileus (Gastrointestinal disorders) | 2 (2) | 1 (1)
Anastomosis leakage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fever (Immune system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No